CLINICAL TRIAL: NCT01641718
Title: Use of Human Fibrin Glue (Tisseel) Versus Staples for Mesh Fixation in Laparoscopic Transabdominal Preperitoneal Hernioplasty (TISTA)
Brief Title: Use of Human Fibrin Glue Versus Staples for Mesh Fixation in Laparoscopic Transabdominal Preperitoneal Hernioplasty
Acronym: TISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sascha Müller (Other)
Responsible Party: Sponsor-Investigator, Sascha Müller, Oberarzt (attending physician), Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TISTA
Record Dates: First submitted 2012-06-29; First posted 2012-07-17 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Hernia, Inguinal
Keywords: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal | interventions — Fibrin Tissue Adhesive; Sutures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single sided glue (Experimental): Mesh is fixed with Tisseel for single sided inguinal hernias.
  Interventions: Drug: Tissue glue
- Single sided stapled (Active Comparator): Mesh is fixed with staples for single sided inguinal hernias.
  Interventions: Device: Staples
- Bilateral glue right (Other): For bilateral inguinal hernias mesh on the right side is fixed with Tisseel, on the left with staples.
  Experimental treatment and active comparator in the same patient.
  Interventions: Drug: Tissue glue; Device: Staples
- Bilateral glue left (Other): For bilateral inguinal hernias mesh on the left side is fixed with Tisseel, on the right with staples.
  Experimental treatment and active comparator in the same patient.
  Interventions: Drug: Tissue glue; Device: Staples

INTERVENTIONS:
Drug: Tissue glue — The mesh fixation for the transabdominal preperitoneal patch plastic repair will be performed with 2 mL of tissue glue.
  Other Names: Tisseel (Baxter)
  Arms: Bilateral glue left; Bilateral glue right; Single sided glue
Device: Staples — The mesh fixation for the transabdominal preperitoneal patch plastic repair will be performed with ProTack (Covidien) and Securestrap (Ethicon) staples.
  Other Names: ProTack (Covidien); Securestrap (Ethicon)
  Arms: Bilateral glue left; Bilateral glue right; Single sided stapled

SUMMARY:
Inguinal hernia repairs belong to the most common surgical procedures worldwide. Increasingly they are performed using endoscopical techniques (laparoscopy). Many surgeons prefer to cover the hernia gap with a mesh to prevent recurrence. For it, the mesh must be fixed tightly, but tension free. During laparoscopic surgery the mesh is fixed commonly with staples or tissue glue. However, it is not uncommon that staples cause pain at the staple sites while moving. In addition, staples can cause scarring of the abdominal wall leading to chronic pain.

Aim of the study is to provide evidence that mesh fixation with tissue glue causes less postoperative pain compared to fixation with staples.

Patients with unilateral inguinal hernia will be randomized to receive either mesh fixation with tissue glue or staples (ratio 1:1).

Patients with bilateral inguinal hernia will receive mesh fixation with tissue glue on one side and staple fixation on the other side. The side treated with tissue glue will be randomized (ratio 1:1).

DETAILED DESCRIPTION:
______________________________________________

The inguinal hernia is the most common hernia, including 90% of all spontaneous hernias, and the inguinal hernia repair is the most frequently performed procedure in general surgery. In the United States more than 700,000 inguinal hernias are repaired annually and in Germany more than 200,000. The standard method for inguinal hernia repair, originally described by Bassini in 1889, is the closure of the inguinal canal using sutures. Due to the high recurrence rate of this technique, methods using the tension-free implantation of synthetic meshes were established. Furthermore, endoscopic/laparoscopy methods were established, in which the hernia canal is usually approached from the posterior side opposite to the anterior site in the open approach. It is still hotly debated which of these approaches and methods is the best. Among the various posterior techniques using preperitoneal mesh implantation, the transabdominal preperitoneal patch plastic repair (TAPP) and the total extraperitoneal (TEP) repair achieved the highest acceptance. There are many indications for the use of both techniques, but the TAPP is recommended especially for recurrent hernias (after open preperitoneal patch plastic) and difficult hernias (sliding or incarcerated hernias). The advantages of the TAPP are that it is easier to perform, has a better possibility of standardization, and offers the option to perform a diagnostic laparoscopy. Thus, the type of hernia can be assessed immediately on both sides and a bilateral repair can be performed without additional incisions. In general, learning TAPP is easier than TEP. Most randomized studies comparing laparoscopic with open repair found the following results for laparoscopy: reduced postoperative pain, earlier return to work, increased costs, increased operating time, longer learning period, and during the early learning phase an increased recurrence and complication rate. In summary open, mesh-based, tension-free repair remains the standard, but laparoscopic herniorrhaphy, in the hands of adequately trained surgeons, produces excellent results comparable to those of open repair.

Whether patients suffer from postoperative pain depends on many factors like the type of intervention, complications, age, and individual tolerance. In particular the type of mesh fixation employed during hernioplasty has a strong influence on postoperative pain. In a recent review mesh fixation by glue was compared to mesh fixation with staplers during endoscopic inguinal hernia repair (Surg Laparosc Endosc Percutan Tech (2010) 20:205). For the transabdominal preperitoneal patch plastic repair two randomized controlled trials, one non randomized trial and two case series were identified in this review. Although the authors found reduced postoperative pain and faster recovery after glue fixation without any significant difference in the recurrence rate, the authors still concluded: "As the overall quality of published data remains poor, further well-designed studies are needed until fibrin sealing can replace mechanical stapling as a new standard for mesh fixation." Thus well designed randomized studies comparing glue vs. staples fixation during TAPP are still warranted. Most of the previous studies applied only one mesh fixation method for patients with bilateral hernias. Only one study compared glue and stapler fixation in single patients with bilateral hernias. In this study a 2x2 design will be used, to compare the two fixation methods in patients with unilateral hernia as well as to compare the two methods in the same patient with bilateral hernias, eliminating the interindividual bias of the single hernia group. Furthermore this study focuses on the early postoperative pain, with a rather thorough coverage in the first 2 days. In many other studies the first time pain is measured is one month after surgery, which is the last time point in this study.

The main aim of this trial is to investigate the early postoperative pain after laparoscopic hernia repair in TAPP technique using either fibrin glue or staples for mesh fixation.

ELIGIBILITY:
Inclusion Criteria:

* primary hernia repair (no re-operation for recurrent hernia)
* good compliance can be expected
* informed consent

Exclusion Criteria:

* chronic pain
* acute pain requiring analgesic others than paracetamol or more than a single dose non-steroidal anti-inflammatory drugs treatment within 48 h before surgery
* current treatment with psychopharmaceutical drugs
* mental incapacity
* known incompatibility (allergies) with the Tisseel compounds

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain after physical stress | 24 h after surgery
  Patient rates his pain on a scale from 0 to 10 (10 equals worst pain imaginable). (NRS numeric rating scale).
  Patient will be asked to bend the hip joint for 90° on the operated side (both sides for patients with bilateral hernia). Then they are asked for the pain rating (physical stress measurement).

SECONDARY OUTCOMES:
Pain at rest | 4, 8, 16, 24, 32, 48 h & 1 month after surgery
  Patient rates his pain on a scale from 0 to 10 (10 equals worst pain imaginable). (NRS numeric rating scale).
  Patient is interviewed for pain at rest before pain measurement after physical stress.
Pain after physical stress | 4, 8, 16, 32, 48 h & 1 month after surgery
  Patient rates his pain on a scale from 0 to 10 (10 equals worst pain imaginable). (NRS numeric rating scale).
  Patient will be asked to bend the hip joint for 90° on the operated side (both sides for patients with bilateral hernia). Then they are asked for the pain rating (physical stress measurement).
Operating time | 4 h
  Time in minutes from the first skin incision to the application of dressing.
Length of hospital stay | 2 weeks
  Time in days (with one decimal) from start of surgery to hospital release.
Postoperative analgetic requirements | 1 month
  Amount (g/day) and type (paracetamol, metamizol, morphin) of analgesic required after surgery until hospital discharge.
Incidence of persisting pain (neuralgia) | 1 month
  Persisting pain (neuralgia) is defined by the presence of intermittent hyperesthesia, burning sensation or jabbing pain in the ipsilateral inguinal area nerves (genitofemoral nerve, lateral cutaneous femoral nerve, ilioinguinal and iliohypogastric nerve).
  Evaluation for chronic pain (neuralgia) will be performed during the 1 month follow-up visit. The degree of pain will measured as described above.
Postoperative morbidity | 1 month
  * Wound infection (defined as those treated without further surgery and identified by clinical examination without microbiological confirmation)
  * haematoma or seroma formation (identified by clinical examination alone before discharge from hospital, without the requirement for radiological confirmation)
  * Re-operation (Need for re-operation during patients' initial hospital stay)
  * Bleeding
  * Urinary retention, urinary tract infection
  * Pulmonary infection
  * Any serious deviation from the normal postoperative course
Medical leave of absence | 2 months
  Time in days from hospital discharge to first working day. All patients will be encouraged to return to work as soon as possible, irrespective of their profession. Time to return to work will be obtained during 1 month follow-up visit. If still on medical leave of absence at this time, patients will be later contacted by phone to obtain the day of return to work. Depending on the expected course of recovery these calls will be performed in a weekly or biweekly fashion.
Economic impact | 2 months
  Will be calculated using the following factors:
  * Cost for glue, staples and instruments to apply glue or staples
  * If relevant: cost for increased operating time for the "slower" mesh fixation technique
  * length of hospital stay (cost/day)
  * medical leave of absence (converted into a monetary amount using an average salary)

CONTACTS AND LOCATIONS:
Overall Officials: Sascha A Müller, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St.Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Muller SA, Warschkow R, Beutner U, Luthi C, Ukegjini K, Schmied BM, Tarantino I. Use of human fibrin glue (Tisseel) versus staples for mesh fixation in laparoscopic transabdominal preperitoneal hernioplasty (TISTA): a randomized controlled trial (NCT01641718). BMC Surg. 2014 Apr 1;14:18. doi: 10.1186/1471-2482-14-18. PMID 24690207
- See also: Website of the Department of Surgery, Cantonal Hospital St. Gallen (German only) — http://www.chirurgie.kssg.ch/home/unsere_klinik.html